CLINICAL TRIAL: NCT02304731
Title: Physical Exercise and Pollution: Cardiorrespiratory, Cerebral and Molecular Aspects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciana Caxa, Master Degree, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UFSao Paulo
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cognitive Function 1, Social
Keywords: Physical Exercise, Atmospheric Pollution, Cognition.
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise and Pollution Groups (Experimental): Physical Exercise performed in a clean environment and in a polluted environment.
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Physical Exercise — Incremental running

SUMMARY:
Modern society increasingly seeks healthy life style, and regular physical activity is considered one of the main factors that improve the quality of life. The evidence shows that the aerobic physical training in controlled environments benefit various aspects of human health, including cognition in the elderly population. However, when exercise is performed in a polluted environment, the individual is subjected to grater exposure to pollutants due to increased ventilation (breathing).

DETAILED DESCRIPTION:
Modern society increasingly seeks healthy life style, and regular physical activity is considered one of the main factors that improve the quality of life. The evidence shows that the aerobic physical training in controlled environments benefit various aspects of human health, including cognition in the elderly population. However, when exercise is performed in a polluted environment, the individual is subjected to grater exposure to pollutants due to increased ventilation (breathing). It is well known that inhaled pollutants can cause oxidative modification in biomolecules and oxidative stress is a cause of diverse diseases. This scenario raises important questions: the deleterious effects of pollution can abolish the beneficial effects of exercise? This issue is currently relevant given the increasing level of air pollution in large urban centers such as Sao Paulo city and at the same time, outdoor physical activity in public places is largely stimulated by public organizations, particularly for elderly. Thus this multidisciplinary project aims to investigate the deleterious effects of urban air pollution in elderly people who practice aerobic physical exercise outdoors in Sao Paulo and compare with those who practice in Laboratory. This study can provide important knowledge for public health and welfare of the population.

ELIGIBILITY:
Inclusion Criteria: Health Subjects that lives in São Paulo city for at least 10 years.

-

Exclusion Criteria: Neuropsychological issues.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cognitive Benefits | 12 weeks
  Neuropsychological Tests applied at the beginning and at the end of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Caxá, Master, Study Chair — Federal University of São Paulo